CLINICAL TRIAL: NCT00129376
Title: Multicenter Phase II Trial of Doxorubicin and Cyclophosphamide (AC) Followed by Weekly Docetaxel (T) as Neoadjuvant Treatment for Operable Stage II and IIIA Breast Cancer Patients
Brief Title: Doxorubicin and Cyclophosphamide (AC) Followed by Weekly Docetaxel as Neoadjuvant Treatment of Breast Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spanish Breast Cancer Research Group (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEICAM 2002-03
Record Dates: First submitted 2005-08-10; First posted 2005-08-11 (Estimated); Results first posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-04

CONDITIONS: Breast Cancer
Keywords: Stage II and IIIA breast Cancer.; Neoadjuvant chemotherapy.; Weekly docetaxel.
MeSH Terms: conditions — Breast Neoplasms | interventions — Doxorubicin; Cyclophosphamide; Docetaxel

ARMS (1):
- Doxorubicin+cyclophosphamide - Docetaxel (Experimental): Patients received doxorubicin (60 mg/m2) and cyclophosphamide (600 mg/m2), both in a short intravenous infusion, every three weeks for four cycles. Later, docetaxel (36 mg/m2) was administered an intravenous infusion, weekly for six weeks followed by a 2-week resting period (8-week cycle).
  Interventions: Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Docetaxel

INTERVENTIONS:
Drug: Doxorubicin
  Other Names: adriamycin
Drug: Cyclophosphamide
  Other Names: Cytoxan
Drug: Docetaxel
  Other Names: Taxotere

SUMMARY:
Treatment consists of 4 AC cycles followed by 2 weekly docetaxel cycles (12 infusions).

The pathological complete response rate obtained in previous studies is around 12%. The expected pathological complete response rate in this study is 25%. With an alpha error of 0.05 and a beta error of 0.2, and following Simon´s 2 phase test, 19 patients are needed initially. With 2 pathological complete responses, patient recruitment will continue until approximately 61 patients are recruited. Twelve pathological complete responses are needed to confirm the study hypothesis.

DETAILED DESCRIPTION:
Patients received doxorubicin (60 mg/m2) and cyclophosphamide (600 mg/m2), both in a short intravenous infusion, every three weeks for four cycles (days 1, 22, 43 and 64). Three weeks later, docetaxel (36 mg/m2) was administered as a 30-min intravenous infusion, weekly for six weeks (days 85, 92, 99, 106, 113 and 120) followed by a 2-week resting period (8-week cycle). After that, patients received a second docetaxel cycle (infusions on days 141, 148, 155, 162, 169 and 176). Adjuvant chemotherapy and radiotherapy were delivered according to the protocol of each participating center. Hormonal treatment was started after the last chemotherapy infusion in all patients with positive estrogen and/or progesterone receptor tumors and was continued for five years.

Semiquantitative determination of three molecular markers was carried out by immunocytochemical methods. Tissue samples were taken prior to initiation of chemotherapy from the core of the primary tumors. Specimens were sent to a central laboratory for analysis of Topo II, survivin and p27.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Patients with breast cancer stages II and IIIA, with histological diagnoses as per true-cut or open biopsy.
* Negative extension study, including bilateral mammography, thoracic x-ray, computed tomography (CT)-scan or abdominal echography and bone scintigraphy.
* Analysis of hormone receptor status in primary tumour. It is highly recommended to obtain a tumour tissue sample before start of treatment, and after definitive surgery. These samples will be analysed centrally by Spanish Breast Cancer Research Group (GEICAM).
* Age >= 18 and <= 70 years old.
* Performance status as per Karnofsky index >= 80.
* Minimum life expectancy of 6 months.
* Electrocardiogram (EKG) 12 weeks before registration to the study. If abnormalities are suspected, cardiac function must be assessed by left ventricular ejection fraction (LVEF).
* Haematology: neutrophils >= 2.0 x10^9/l; platelets >= 100 x10^9/l; hemoglobin >=10 g/dl.
* Hepatic function: total bilirubin <= 1 x upper normal limit (UNL); Aspartate aminotransferase (AST) (SGOT) and and Alanine aminotransferase (ALT) (SGPT) <= 2.5 x UNL; alkaline phosphatase <= 5 x UNL.
* Renal function: creatinine <= 1.5 x UNL; creatinine clearance >= 60 ml/min.
* Patients able to comply with study requirements.
* Negative pregnancy test.
* Adequate contraceptive method during the study and up to 3 months after definitive surgery.

Exclusion Criteria:

* Previous systemic therapy for breast cancer treatment.
* Previous treatments with anthracyclines or taxanes for any malignancy.
* Previous radiotherapy for breast cancer.
* Bilateral invasive breast cancer.
* Pregnant or lactating women.
* Previous motor or sensorial neurotoxicity grade >=2.
* Other serious pathologies: congestive heart failure or angina pectoris; history of myocardial infarction in the previous year; uncontrolled hypertension (HT) or high risk arrhythmias.
* History of neurological or psychiatric impairment, precluding patients from providing free informed consent.
* Active infection.
* Active peptic ulcer; unstable diabetes mellitus.
* History of previous or current malignancies other than breast cancer, except for basal skin carcinoma, cervical in situ carcinoma, other tumour diagnosed and treated more than 10 years before, ductal carcinoma in situ (DCIS) or lobular carcinoma in situ (LCIS).
* Chronic treatment with corticoids unless the treatment started > 6 months before registration to the study, and low doses are administered.
* Substitutive hormonal therapy. This treatment must be interrupted before inclusion in the study.
* Concomitant treatment with other investigational products or administration in the 30 previous days.
* Males.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2003-02 (Actual); Primary Completion 2005-07 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz; Study Director, Study Director — Hospital Universitario Marqués de Valdecilla
Locations (6):
- Spain (6):
  - Hospital Universitario Germans Trias i Pujol, Badalona, Barcelona
  - Corporació Sanitaria Parc Taulí, Sabadell, Barcelona
  - Hospital de la Ribera, Alzira, Valencia
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital General Universitario de Alicante, Alicante
  - Fundación Jiménez Díaz, Madrid

REFERENCES:
- See also: Click here for more information about this study: GEICAM 2002-03 — http://www.geicam.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Doxorubicin + Cyclophosphamide Followed Docetaxel: Patients received doxorubicin (60 mg/m2) and cyclophosphamide (600 mg/m2), both in a short intravenous infusion, every three weeks for four cycles (days 1, 22, 43 and 64). Three weeks later, docetaxel (36 mg/m2) was administered as a 30-min intravenous infusion, weekly for six weeks (days 85, 92, 99, 106, 113 and 120) followed by a 2-week resting period (8-week cycle). After that, patients received a second docetaxel cycle (infusions on days 141, 148, 155, 162, 169 and 176).
Period: Overall Study
Arm/Group | Doxorubicin + Cyclophosphamide Followed Docetaxel
Started | 63
Completed | 61
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Doxorubicin + Cyclophosphamide Followed Docetaxel
Number analyzed (Participants) | 63
Age, Continuous [Median (Full Range); unit: years] | 48.43 [25 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 63
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Spain | 63
Menopausal status [Count of Participants; unit: Participants]
  Premenopausal | 35
  Postmenopausal | 28
Median Tumor size, cm [Median (Full Range); unit: cm] | 4.8 [2.0 to 12.5]
Disease stage (I, IIA, IIB y IIIA) [Count of Participants; unit: Participants] — Stage was classified following the TNM system of the American Joint Committee on Cancer (AJCC).
  Stage 0. Cancer in situ ("in place"). Still located in the place they started and have not spread to nearby tissues. This stage is highly curable, by removing the entire tumor with surgery.
  Stage I. Small cancer that has not grown into nearby tissues. Also has not spread.
  Stage II and Stage III. Larger cancers that have grown deeply into nearby tissue. They may have also spread to lymph nodes but not to other parts of the body.
  Stage IV. Cancer has spread to other organs or parts of the body.
  Participants
    I | 1
    IIA | 23
    IIB | 35
    IIIA | 4
Hormonal receptors (Estrogen Receptor [ER]+/ Progesterone Receptor [PR]+, ER+/PR-, ER-/PR+, ER-/PR-) [Count of Participants; unit: Participants]
  ER+/PR+ | 32
  ER+/PR- | 18
  ER-/PR+ | 3
  ER-/PR- | 10

OUTCOME MEASURES:

1. Primary Outcome: Pathological Complete Response (pCR) Rate
Description: Pathological complete response was defined by the Miller & Payne criteria. pCR was defined as no invasive cells identifiable in breast sections at surgery. Response was measured by physical exam and breast imaging before surgery and was evaluated according to the World Health Organization (WHO) criteria. Pathological response after surgery, was based on the proportion of remaining tumor and postchemotherapy changes, evaluating separately the response in the breast and in the axilla lymph nodes.
Time Frame: Up to 29 weeks
Population: 2 patients did not received surgery, 1 because of disease progression, and 1 due to inacceptable toxicity.
Measure: Count of Participants; unit: Participants
Arm/Group | Doxorubicin + Cyclophosphamide Followed Docetaxel
Number analyzed (Participants) | 61
Participants | 11

2. Secondary Outcome: Clinical Response Rate (CRR)
Description: CRR measured according to the Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions, where:
  * Complete Response (CR): disappearance of all target lesions
  * Partial Response (PR): >=30% decrease in the sum of the longest diameter of target lesions
  * Progresive Disease (PD): >=20% increase from smallest sum of longest diameter recorded since treatment started (best response).
  * Stable Disease (SD): Neither PD nor PR
Time Frame: Up to 29 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Doxorubicin + Cyclophosphamide Followed Docetaxel
Number analyzed (Participants) | 63
Participants
  Complete response | 29
  Partial response | 28
  Stable Disease | 5
  Unknown | 1

3. Secondary Outcome: Number of Participants With Over-expression of Topo II (>10% Cells With Nuclear Staining)
Description: Paraffin-embedded tumors were processed with standard immunocytochemical techniques. Over-expression of Topo II was defined as >10% cells with nuclear staining.
Time Frame: Up to 29 weeks
Population: 20 patient tumor sample could not be evaluated
Measure: Count of Participants; unit: Participants
Arm/Group | Doxorubicin + Cyclophosphamide Followed Docetaxel
Number analyzed (Participants) | 41
Participants
  > 10% | 20
  < 10% | 21

4. Secondary Outcome: Number of Participants With Over-expression of Survivin (>1% Cells With Nuclear Staining)
Description: Paraffin-embedded tumors were processed with standard immunocytochemical techniques. Tumors with more than 1% of cells with nuclear staining were considered to be over-expressing this protein.
Time Frame: Up to 29 weeks
Population: 17 patient tumor sample could not be evaluated
Measure: Count of Participants; unit: Participants
Arm/Group | Doxorubicin + Cyclophosphamide Followed Docetaxel
Number analyzed (Participants) | 44
Participants
  > 1 % | 18
  < 1% | 26

5. Secondary Outcome: Number of Participants With Over-expression of p27 (>75% Cells With Nuclear Staining)
Description: Paraffin-embedded tumors were processed with standard immunocytochemical techniques. Sections were rated according to the percentage of tumor cells nuclei with positive staining (1 = < 25%; 2 = between 25-75% and 3 = > 75%).
Time Frame: Up to 29 weeks
Population: 20 patient tumor sample could not be evaluated
Measure: Count of Participants; unit: Participants
Arm/Group | Doxorubicin + Cyclophosphamide Followed Docetaxel
Number analyzed (Participants) | 41
Participants
  < 75% | 24
  > 75% | 17

ADVERSE EVENTS:
Time Frame: Through study treatment up to surgery, an average of 26 weeks
Arm/Group | Doxorubicin + Cyclophosphamide Followed Docetaxel
All-Cause Mortality (participants affected / at risk) | 0/63
Serious Adverse Events (participants affected / at risk) | 12/63
Other Adverse Events (participants affected / at risk) | 63/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Doxorubicin + Cyclophosphamide Followed Docetaxel (N=63)
Acute Pharyngitis (Infections and infestations) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (4) — Grade 3
Neutrophil count decreased (Investigations) | 1 (1) — Grade 3
Infection (Infections and infestations) | 3 (3)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Grade 2
Vomiting (Gastrointestinal disorders) | 1 (1) — Grade 3
Congestive heart failure (Cardiac disorders) | 1 (1) — Left Ventricular Ejection Fraction Grade 4
Cardiac-ischemia/infarction (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Doxorubicin + Cyclophosphamide Followed Docetaxel (N=63)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 — Grade 3
Leukopenia (Blood and lymphatic system disorders) | 5 — Grade 3
Lymphopenia (Blood and lymphatic system disorders) | 26 — Grade 4
Neutropenia (Blood and lymphatic system disorders) | 10 — Grade 3
Anxiety (Nervous system disorders) | 1 — Grade 3
Congestive heart failure (Cardiac disorders) | 1 — Grade 3
Diarrhoea (Gastrointestinal disorders) | 1 — Grade 3
Dry skin (Skin and subcutaneous tissue disorders) | 1 — Grade 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 — Grade 4
Edema (Cardiac disorders) | 1 — Grade 3
Asthenia (General disorders) | 5 — Grade 3
Hepatic dysfunction (Hepatobiliary disorders) | 2 — Grade 3
Infection without neutropenia (Infections and infestations) | 1 — Grade 3
Nausea (Gastrointestinal disorders) | 2 — Grade 3
Syncope (Nervous system disorders) | 1 — Grade 3
Vomiting (Gastrointestinal disorders) | 5 — Grade 3
Weight loss (General disorders) | 1 — Grade 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less